CLINICAL TRIAL: NCT06882447
Title: A Prospective, Single-center, Single-arm, Phase II Study of QL1706 Combined with Nine价HPV Vaccine As First-line Treatment for Persistent, Recurrent or Metastatic Cervical Cancer
Brief Title: A Study of QL1706 Combined with Nine HPV Vaccine As First-line Treatment for Persistent, Recurrent or Metastatic Cervical Cancer
Acronym: QL1706
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Buhai Wang, Chief of Oncology, Northern Jiangsu People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ky030
Record Dates: First submitted 2025-03-04; First posted 2025-03-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer Stage IVB
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Other): Trial drug: QL1706, HPV 9-valent vaccine
  Interventions: Drug: Trial drug: QL1706, HPV 9-valent vaccine

INTERVENTIONS:
Drug: Trial drug: QL1706, HPV 9-valent vaccine — QL1706: Dose: 5 mg/kg ; intravenous infusion (ivgtt), administered on day 1 of each cycle and once every 3 weeks (21 days).

SUMMARY:
The study medications were used as follows: 1 cycle every 21 days (3 weeks) of the following regimen.

Test drug: QL1706, HPV 9-valent vaccine

QL1706: Dose: 5 mg/kg ; intravenous infusion (ivgtt), administered on Day 1 of each cycle and every 3 weeks (21 days).

Treatment will continue until loss of clinical benefit, occurrence of intolerable toxicity, patient or physician decision to discontinue treatment, death of the patient receiving the experimental treatment, or completion of 2 years of dosing (35 dosing cycles), withdrawal of informed consent by the subject, pregnancy of the subject, noncompliance with protocol or procedural requirements, or for administrative reasons.

HPV 9-valent vaccine: 1st dose 1 day prior to first QL1706 administration; 2nd dose 2 months after 1st dose; 3rd dose 6 months after 1st dose.

ELIGIBILITY:
1. Patients with unsystematically treated cervical cancer, who voluntarily participate in the clinical study; fully understand and informed about the study and sign the Informed Consent Form (ICF); willing to follow and have the ability to complete all the trial procedures.
2. With histologically confirmed diagnosis of cervical cancer, a pathology report and pathology slides are required.
3. have at least one measurable lesion as assessed by the investigator according to RECIST 1.1.

   Note: Measurable target lesions cannot be selected from previous radiotherapy sites. If the target lesion at the site of prior radiotherapy is the only optional target lesion, the investigator is required to provide anterior and posterior imaging data showing significant progression of this lesion.
4. Recovery of AE associated with prior antitumor therapy to CTCAE ≤ Grade 1 (except for Grade 2 alopecia).
5. ECOG score ≤ 1 within 7 days prior to first dose of study drug.
6. expected survival ≥ 12 weeks.
7. Subjects with chronic HBV infection must have HBV-DNA < 1000 copies/ml and must agree to receive antiviral therapy according to treatment guidelines for patients with hepatitis B surface antigen positivity; patients with HCV-RNA positivity must agree to receive antiviral therapy according to treatment guidelines and have liver function at CTCAE ≤ grade 1.
8. Normal major organ function, i.e., the following criteria are met (no transfusion, erythropoietin, or colony-stimulating factor (G-CSF) therapy within 14 days prior to administration of study drug) Hematologic Neutrophils (ANC) ≥ 1.5 x 109/L Platelets (PLT) ≥ 90×109/L Hemoglobin (Hb) ≥ 90g/L Liver Function Total bilirubin (TBIL) ≤ 1.5 x upper limit of normal (ULN) Glutamate aminotransferase (ALT) ≤ 2.5×ULN; For patients with liver metastases ≤ 5 × ULN Aspartate aminotransferase (AST) ≤ 2.5 × ULN; For patients with liver metastases ≤ 5×ULN Renal Function Creatinine (Cr) ≤ 1.5×ULN; If > 1.5 x ULN, creatinine clearance ≥ 50 ml/min. (calculated according to the Cockcroft-Gault formula) Coagulation Activated partial thromboplastin time (APTT) ≤ 1.5 x ULN Prothrombin time (PT) ≤ 1.5×ULN International normalized ratio (INR) ≤ 1.5×ULN
9. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to initiation of study drug and be willing to use a hi ghly effective method of contraception for the duration of the trial and for 90 days after the last administration of the test drug.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
orr | every 6 weeks (±7 days)
  Evaluating the objective remission rate (ORR) of QL1706 in combination with the nine-valent HPV vaccine for the first-line treatment of persistent, recurrent or metastatic cervical cancer